CLINICAL TRIAL: NCT02209818
Title: Evaluation of Low Level Laser Therapy (LLLT) Effect on Pain Management Caused by Orthodontic Elastomeric Separators
Brief Title: Effect of Laser Application in Pain Management Following the Use of Orthodontic Elastomeric Separators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Perio-06-2014
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Orthodontic Treatment
Keywords: Low level laser therapy; Elastomeric separator; Placebo; Visual analog scale; Laser irradiation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser Irradiation One Dose (Experimental): Laser irradiation will be applied in one dose for patients in this group, but only on one side of the jaw. The other side of the jaw will receive a placebo procedure (i.e. a red light beam will be emitted on the gingival tissues as if they are irradiated by a laser beam).
  Interventions: Radiation: Laser Irradiation One dose
- Laser Irradiation Two doses (Experimental): Laser irradiation will be applied in two doses for patients in this group, but only on one side of the jaw. The second dose will be given after 24 hour of the first one. The other side of the jaw will receive a placebo procedure (i.e. a red light beam will be emitted on the gingival tissues as if they are irradiated by a laser beam).
  Interventions: Radiation: Laser Irradiation Two doses

INTERVENTIONS:
Radiation: Laser Irradiation One dose
  Arms: Laser Irradiation One Dose
Radiation: Laser Irradiation Two doses
  Arms: Laser Irradiation Two doses

SUMMARY:
The aim of this study is to evaluate the effect of low level laser therapy (LLLT) on pain management in people commencing orthodontic treatment. The study design is a randomized controlled trial.

Participants' pain will be dealt with by laser irradiation in one side of the jaw randomly, and the other side will be treated by a placebo procedure. Pain assessment will be measured using Visual Analog Scales (VAS).

The hypothesis of this study is that laser irradiation decreases the amount of pain following the insertion of orthodontic separators.

DETAILED DESCRIPTION:
Here we have two groups:

The first group will undergo one dose of irradiation which is going to be applied on one side of the mouth whereas the opposing side will serve as a control side (placebo).

The second group will undergo two doses of irradiation which is going to be applied on one side of the mouth whereas the opposing side will serve as a control side (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Participants should have healthy periodontal structures, healthy teeth.
* Presence of first molar in both side of the jaw.

Exclusion Criteria:

* systemic diseases
* chronic pain or neurological pain

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Pain Perception | Pain will be evaluated at 1, 6, 24, 48, and 72 hours after laser irradiation
  Pain assessment will be performed using a Visual Analog Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Mai Almallah, DDS, Principal Investigator — MSc student, Department of Periodontics, University of Damascus Dental School, Damascus; Mohammad Y Hajeer, DDS MSc PhD, Study Director — Associate Professor, Orthodontics Department, University of Damascus Dental School, Damascus; Wael Mahdi, DDS MSc PhD, Study Director — Senior Lecturer in Periodontics, Periodontics Department, University of Damascus Dental School
Locations (1):
- Department of Periodontics, University of Damascus Dental School, Damascus, Rif-dimashq Governorate, Syria

REFERENCES:
- [Background] Abtahi SM, Mousavi SA, Shafaee H, Tanbakuchi B. Effect of low-level laser therapy on dental pain induced by separator force in orthodontic treatment. Dent Res J (Isfahan). 2013 Sep;10(5):647-51. PMID 24348624
- [Background] Eslamian L, Borzabadi-Farahani A, Hassanzadeh-Azhiri A, Badiee MR, Fekrazad R. The effect of 810-nm low-level laser therapy on pain caused by orthodontic elastomeric separators. Lasers Med Sci. 2014 Mar;29(2):559-64. doi: 10.1007/s10103-012-1258-1. Epub 2013 Jan 20. PMID 23334785
- [Background] Nobrega C, da Silva EM, de Macedo CR. Low-level laser therapy for treatment of pain associated with orthodontic elastomeric separator placement: a placebo-controlled randomized double-blind clinical trial. Photomed Laser Surg. 2013 Jan;31(1):10-6. doi: 10.1089/pho.2012.3338. Epub 2012 Nov 15. PMID 23153291
- [Background] Artes-Ribas M, Arnabat-Dominguez J, Puigdollers A. Analgesic effect of a low-level laser therapy (830 nm) in early orthodontic treatment. Lasers Med Sci. 2013 Jan;28(1):335-41. doi: 10.1007/s10103-012-1135-y. Epub 2012 Jul 21. PMID 22814893
- [Background] Huang TH, Liu SL, Chen CL, Shie MY, Kao CT. Low-level laser effects on simulated orthodontic tension side periodontal ligament cells. Photomed Laser Surg. 2013 Feb;31(2):72-7. doi: 10.1089/pho.2012.3359. Epub 2013 Jan 17. PMID 23327633
- [Background] Kim WT, Bayome M, Park JB, Park JH, Baek SH, Kook YA. Effect of frequent laser irradiation on orthodontic pain. A single-blind randomized clinical trial. Angle Orthod. 2013 Jul;83(4):611-6. doi: 10.2319/082012-665.1. Epub 2012 Dec 14. PMID 23241006
- [Background] Fujiyama K, Deguchi T, Murakami T, Fujii A, Kushima K, Takano-Yamamoto T. Clinical effect of CO(2) laser in reducing pain in orthodontics. Angle Orthod. 2008 Mar;78(2):299-303. doi: 10.2319/033007-153.1. PMID 18251609